CLINICAL TRIAL: NCT07332169
Title: The Efficacy of Non-invasive Brain Stimulation on Cognitive Functions in Patients With Chronic Obstructive Pulmonary Disease: Double-Blinded Randomised Controlled Trial
Acronym: NIBS COPD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shahad Abdulrahman Alkandari (Other Government)
Collaborators: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Sponsor-Investigator, Shahad Abdulrahman Alkandari, Shahad Alkandari MSc, PT., Ministry of Health, Kuwait
Organization: Ministry of Health, Kuwait (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-PGS-2025-03-0600; IRB-PGS-2025-03-0553 (Other: Imam Abdulrahman Bin Faisal University)
Record Dates: First submitted 2025-12-28; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: COPD; COPD (Chronic Obstructive Pulmonary Disease); Cognitive Impairment (CI); Non-invasive Brain Stimulation
Keywords: COPD; NIBS; non-invasive brain stimulation; cognitive function; cognitive impairment
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Two groups included: One group will receive the non-invasive brain stimulation, and the other group will receive sham non-invasive brain stimulation.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-invasive brain stimulation (Experimental): Sinusoidal current used between two electrodes on the dorsolateral prefrontal cortex (DLPFC) area. - Gamma-Transcranial Alternating Current Stimulation (tACS) of 2 mA at 40 Hz will be given to the experimental group. - Session duration will last 20 minutes, of 5 session/week, for 3weeks.
  Interventions: Device: Non-invasive brain stimulation
- Sham Non-invasive brain stimulation (Sham Comparator): Sinusoidal current used between two electrodes on the dorsolateral prefrontal cortex (DLPFC) area. - To maintain this stimulation's indistinguishability from the experimental stimulation, the control group will be given an electric current that ramps down 60 seconds after the stimulation begins. - Session duration will last 20 minutes, of 5 session/week, for 3weeks.
  Interventions: Device: Sham Non-Invasive brain stimulation

INTERVENTIONS:
Device: Non-invasive brain stimulation — Non-invasive brain stimulation (NIBS) modifies brain activity without surgery using electric currents. - Transcranial alternating current stimulation (tACS) is one type of NIBS that modifies neuronal oscillations in the brain by applying alternating electrical currents to the scalp through electrodes. - This method can enhance motor abilities, improve cognitive functions, and be used in rehabilitation. - It does this by entraining neurones, which synchronise their firing to the applied sinusoidal frequency. Gamma-Transcranial Alternating Current Stimulation (tACS) of 2 mA at 40 Hz will be given to the experimental group.
  Other Names: NIBS
  Arms: Non-invasive brain stimulation
Device: Sham Non-Invasive brain stimulation — Non-invasive brain stimulation (NIBS) modifies brain activity without surgery using electric currents. - Transcranial alternating current stimulation (tACS) is one type of NIBS that modifies neuronal oscillations in the brain by applying alternating electrical currents to the scalp through electrodes. - This method can enhance motor abilities, improve cognitive functions, and be used in rehabilitation. - It does this by entraining neurones, which synchronise their firing to the applied sinusoidal frequency. The electric current used as ramps down 60 seconds after the stimulation begins.
  Other Names: NIBS
  Arms: Sham Non-invasive brain stimulation

SUMMARY:
The goal of this clinical trial is to examine if non-invasive brain stimulation (NIBS) can enhance cognitive function with chronic obstructive pulmonary disease (COPD) population. The main questions it aims to answer are:

* What is the possibility effect of using the NIBS on cognitive functions as well as the cardiopulmonary parameters in COPD population?
* What is the relation between cognitive function parameters and cardiopulmonary parameters in COPD population who suffer from cognitive impairment (CI)? Researchers will compare NIBS to a sham-NIBS to see if NIBS works to improve cognitive function in COPD population.

Participants will:

Receive NIBS or a sham-NIBS 5 sessions/week for 3 weeks for 20 min each session.

Visit the clinic at the beginning for baseline assessment then after the completion of the 3 weeks to reassess them.

Outcome measures for cognitive parameters and pulmonary parameters will be taken pre and post NIBS intervention

DETAILED DESCRIPTION:
* With over 3.2 million fatalities worldwide, chronic obstructive pulmonary disease (COPD) is considered the third most common cause of mortality and a potentially fatal illness.
* Due to anomalies in the lung architecture, COPD is characterised by a variety of respiratory symptoms.
* Cognitive impairment (CI) is one of the problems caused by COPD that extends beyond the respiratory system.
* The quality of life, treatment compliance, and declines in the condition of COPD patients were all negatively impacted by CI.
* As of right now, no intervention has been promised to improve CI in patients with COPD.

Objective:

To find out how well non-invasive brain stimulation (NIBS), a novel technique, affects cognitive performance in COPD patients

Methods:

* Both the participants and the outcome assessor will be in a double-blind RCT.
* King Fahad University Hospital will be the source of the entirely voluntary participants.
* The IRB of the Imam Abdulrahman bin Faisal institutions accepted the study protocol.
* Following an evaluation using the Montreal Cognitive Assessment Test (MoCA), participants will be divided into four groups based on GOLD: mild GOLD 1, moderate GOLD 2, severe GOLD 3, and very severe GOLD 4.
* For three weeks, both groups will participate in five NIBS sessions per week. While the control group will receive sham brain stimulation, the experimental group will receive active brain stimulation.
* Both groups will undergo the evaluation before and after the treatment sessions.
* Primary outcome measurements are battery cognition tests; secondary measures include ABGs, ultrasonography, and cardiopulmonary exercise tests.
* Independent t-tests will be applied to evaluate the differences between the two groups.
* The study will use a two-way repeated measures Analysis of Variance (ANOVA) to determine the intervention's efficacy.
* The association between the improvement of cognitive function and certain factors will be ascertained via the Pearson correlation coefficient.
* The significance level will be set at a p-value of less than 0.05.

Significant:

* We hope that the findings of this study will serve as a helpful guide when deciding how to improve CI in patients with COPD and enhance the treatment strategy for this group.
* The findings of this study will investigate whether NIBS, which is beneficial in another population, can enhance cognitive function in individuals with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Adult age from eighteen years old and above.
* Patients with confirmed COPD via pulmonary function test (PFT) according to the classifications of GOLD.
* All stages of GOLD will be included
* Stable patients, which means they were not admitted to the hospital in the last 3 months
* Patients with COPD with confirmed cognitive impairment by MoCA test.
* All MoCA stages will be included.

Exclusion Criteria:

* Patients without COPD
* Unstable patients with several admission in the last 3 months
* Patients with COPD but without cognitive impairment.
* COPD patients who suffered from any neurological problems
* COPD patients who are contraindicated for using brain stimulation like psychiatric disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
The battery of neurocognitive tests | At enrolment as baseline assessment and at the end of treatment at 3 weeks
  • Neuropsychological tests are going to be utilised to evaluate cognitive function. • The two key domains to be evaluated are memory and attention. • The Flanker Task will test the attention domain by examining how well the executive control network can be modulated by focusing on one stimulus while concurrently preventing the detection of another stimulus. • The Memory Automaticity Task will be used to evaluate working memory, requiring participants to complete Sternberg-style memory searches in order to attain automaticity; Recalling the existence of a specific letter in the memory set and accurately classifying it are prerequisites for this task. - The previously trained researcher will administer the test.

SECONDARY OUTCOMES:
Cardiopulmonary exercise test (CPET) | At enrolment as baseline assessment and at the end of treatment at 3 weeks
  • The gold standard exercise test for calculating VO2 max is the cardiopulmonary exercise (CPET). • It will be used to evaluate COPD patients' functional capacity and VO2max. Each subject will be assessed using incremental CPET at maximal effort. • The modified Bruce procedure will be used to conduct the test on a treadmill. • Breath-by-breath analysis will be used to evaluate the following gas-exchange and ventilation measurements: VO2, end-tidal pressures for carbon dioxide and oxygen (PETCO2 and PETO2), ventilatory equivalents for carbon dioxide (VE/VCO2), and minute ventilation (VE). - The previously trained researcher will administer the test.
Transcranial Doppler (TCD) ultrasound | At enrolment as baseline assessment and at the end of treatment at 3 weeks
  - Transcranial Doppler (TCD) ultrasound allows for the real-time monitoring of cerebrovascular haemodynamic and blood flow parameters throughout the brain's basal arteries. - Taking into account both the end-diastolic and peak systolic flow velocities, the mean flow velocity (MFV) is calculated, and a few important intracranial arteries are evaluated using the temporal bone window. - Qualified neurologists and vascular technologists will conduct the exam.
Arterial blood gas analysis (ABGs) | At enrolment as baseline assessment and at the end of treatment at 3 weeks
  • The acid-base balance and arterial blood oxygenation are measured by arterial blood gas analysis (ABGs), which uses blood drawn from an artery. • We shall test the arterial carbon dioxide tension (PCO2), arterial blood gas oxygen tension (PO2), and pH. • Patients requiring oxygen will be assessed while using their typical inspiratory oxygen fraction. * The test will be done as part of a hospital's routine.

OTHER OUTCOMES:
Montreal Cognitive Assessment (MoCA) Test | Stratification outcome measure only at the beginning of the study
  * MoCA was employed as a stratification result measure at the start of the enrolment process. * MoCA is used to examine various cognitive areas to detect participants' cognitive impairment (CI). * MoCA test scores range from zero to 30, with a score of more than 26 considered CI. * The previously trained researcher will administer the test.

CONTACTS AND LOCATIONS:
Locations (1):
- Imam Abdulrahman Bin Faisal University, Dammam, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Woods AJ, Antal A, Bikson M, Boggio PS, Brunoni AR, Celnik P, Cohen LG, Fregni F, Herrmann CS, Kappenman ES, Knotkova H, Liebetanz D, Miniussi C, Miranda PC, Paulus W, Priori A, Reato D, Stagg C, Wenderoth N, Nitsche MA. A technical guide to tDCS, and related non-invasive brain stimulation tools. Clin Neurophysiol. 2016 Feb;127(2):1031-1048. doi: 10.1016/j.clinph.2015.11.012. Epub 2015 Nov 22. PMID 26652115
- [Background] Lefaucheur JP, Antal A, Ayache SS, Benninger DH, Brunelin J, Cogiamanian F, Cotelli M, De Ridder D, Ferrucci R, Langguth B, Marangolo P, Mylius V, Nitsche MA, Padberg F, Palm U, Poulet E, Priori A, Rossi S, Schecklmann M, Vanneste S, Ziemann U, Garcia-Larrea L, Paulus W. Evidence-based guidelines on the therapeutic use of transcranial direct current stimulation (tDCS). Clin Neurophysiol. 2017 Jan;128(1):56-92. doi: 10.1016/j.clinph.2016.10.087. Epub 2016 Oct 29. PMID 27866120
- [Background] Antal A, Alekseichuk I, Bikson M, Brockmoller J, Brunoni AR, Chen R, Cohen LG, Dowthwaite G, Ellrich J, Floel A, Fregni F, George MS, Hamilton R, Haueisen J, Herrmann CS, Hummel FC, Lefaucheur JP, Liebetanz D, Loo CK, McCaig CD, Miniussi C, Miranda PC, Moliadze V, Nitsche MA, Nowak R, Padberg F, Pascual-Leone A, Poppendieck W, Priori A, Rossi S, Rossini PM, Rothwell J, Rueger MA, Ruffini G, Schellhorn K, Siebner HR, Ugawa Y, Wexler A, Ziemann U, Hallett M, Paulus W. Low intensity transcranial electric stimulation: Safety, ethical, legal regulatory and application guidelines. Clin Neurophysiol. 2017 Sep;128(9):1774-1809. doi: 10.1016/j.clinph.2017.06.001. Epub 2017 Jun 19. PMID 28709880
- [Background] Manippa V, Palmisano A, Nitsche MA, Filardi M, Vilella D, Logroscino G, Rivolta D. Cognitive and Neuropathophysiological Outcomes of Gamma-tACS in Dementia: A Systematic Review. Neuropsychol Rev. 2024 Mar;34(1):338-361. doi: 10.1007/s11065-023-09589-0. Epub 2023 Mar 6. PMID 36877327
- [Background] Chaieb L, Antal A, Pisoni A, Saiote C, Opitz A, Ambrus GG, Focke N, Paulus W. Safety of 5 kHz tACS. Brain Stimul. 2014 Jan-Feb;7(1):92-6. doi: 10.1016/j.brs.2013.08.004. Epub 2013 Sep 13. PMID 24064065
- [Background] Bikson M, Datta A, Elwassif M. Establishing safety limits for transcranial direct current stimulation. Clin Neurophysiol. 2009 Jun;120(6):1033-4. doi: 10.1016/j.clinph.2009.03.018. Epub 2009 Apr 24. No abstract available. PMID 19394269
- [Background] Zhou D, Li A, Li X, Zhuang W, Liang Y, Zheng CY, Zheng H, Yuan TF. Effects of 40 Hz transcranial alternating current stimulation (tACS) on cognitive functions of patients with Alzheimer's disease: a randomised, double-blind, sham-controlled clinical trial. J Neurol Neurosurg Psychiatry. 2022 May;93(5):568-570. doi: 10.1136/jnnp-2021-326885. Epub 2021 Nov 11. No abstract available. PMID 34764150
- [Background] Antal A, Herrmann CS. Transcranial Alternating Current and Random Noise Stimulation: Possible Mechanisms. Neural Plast. 2016;2016:3616807. doi: 10.1155/2016/3616807. Epub 2016 May 3. PMID 27242932
- [Background] Guerra A, Suppa A, Bologna M, D'Onofrio V, Bianchini E, Brown P, Di Lazzaro V, Berardelli A. Boosting the LTP-like plasticity effect of intermittent theta-burst stimulation using gamma transcranial alternating current stimulation. Brain Stimul. 2018 Jul-Aug;11(4):734-742. doi: 10.1016/j.brs.2018.03.015. Epub 2018 Mar 24. PMID 29615367
- [Background] Antal A, Boros K, Poreisz C, Chaieb L, Terney D, Paulus W. Comparatively weak after-effects of transcranial alternating current stimulation (tACS) on cortical excitability in humans. Brain Stimul. 2008 Apr;1(2):97-105. doi: 10.1016/j.brs.2007.10.001. Epub 2007 Dec 3. PMID 20633376
- [Background] GOLD. Global Strategy for the Diagnosis, Management, and Prevention of Chronic Obstructive Pulmonary Disease 2023 REPOR. 2023.
- [Background] Tahasildar KK, Shrawasti SJ, Shete JS. Study of Arterial Blood Gas Analysis (ABG) in Patients of Obstructive Airway Diseases in Accordance with Clinical Correlation. Res J Med Sci. 2024;18:341-5.
- [Background] Dash M, Apsara N, Chitra A. ABG Analysis and its Interpretation. Acta Scientific Paediatrics. 2019;2(10):108-11.
- [Background] Bonow RH, Young CC, Bass DI, Moore A, Levitt MR. Transcranial Doppler ultrasonography in neurological surgery and neurocritical care. Neurosurg Focus. 2019 Dec 1;47(6):E2. doi: 10.3171/2019.9.FOCUS19611. PMID 31786564
- [Background] Purkayastha S, Sorond F. Transcranial Doppler ultrasound: technique and application. Semin Neurol. 2012 Sep;32(4):411-20. doi: 10.1055/s-0032-1331812. Epub 2013 Jan 29. PMID 23361485
- [Background] Guazzi M, Arena R, Halle M, Piepoli MF, Myers J, Lavie CJ. 2016 Focused Update: Clinical Recommendations for Cardiopulmonary Exercise Testing Data Assessment in Specific Patient Populations. Circulation. 2016 Jun 14;133(24):e694-711. doi: 10.1161/CIR.0000000000000406. Epub 2016 May 2. PMID 27143685
- [Background] Shiffrin R, Schneider W. Controlled and automatic human information processing: II. Perceptual learning, automatic attending and a general theory. Psychological Review. 1977;84:127-90.
- [Background] Diamond A. Executive functions. Annu Rev Psychol. 2013;64:135-68. doi: 10.1146/annurev-psych-113011-143750. Epub 2012 Sep 27. PMID 23020641
- [Background] Nasreddine ZS, Phillips NA, Bédirian V, Charbonneau S, Whitehead V, Collin I, et al. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005;53(4):695-9.
- [Background] Rahman TT, El Gaafary MM. Montreal Cognitive Assessment Arabic version: reliability and validity prevalence of mild cognitive impairment among elderly attending geriatric clubs in Cairo. Geriatr Gerontol Int. 2009 Mar;9(1):54-61. doi: 10.1111/j.1447-0594.2008.00509.x. PMID 19260980
- [Background] Kaya M, Gurses HN, Ucgun H, Okyaltirik F. Effects of creative dance on functional capacity, pulmonary function, balance, and cognition in COPD patients: A randomized controlled trial. Heart Lung. 2023 Mar-Apr;58:13-20. doi: 10.1016/j.hrtlng.2022.10.017. Epub 2022 Nov 3. PMID 36335909
- [Background] Leitao J, Thielscher A, Tunnerhoff J, Noppeney U. Concurrent TMS-fMRI Reveals Interactions between Dorsal and Ventral Attentional Systems. J Neurosci. 2015 Aug 12;35(32):11445-57. doi: 10.1523/JNEUROSCI.0939-15.2015. PMID 26269649
- [Background] Hsueh JJ, Chen TS, Chen JJ, Shaw FZ. Neurofeedback training of EEG alpha rhythm enhances episodic and working memory. Hum Brain Mapp. 2016 Jul;37(7):2662-75. doi: 10.1002/hbm.23201. Epub 2016 Apr 1. PMID 27038114
- [Background] Shen J, Zhang G, Yao L, Zhao X. Real-time fMRI training-induced changes in regional connectivity mediating verbal working memory behavioral performance. Neuroscience. 2015 Mar 19;289:144-52. doi: 10.1016/j.neuroscience.2014.12.071. Epub 2015 Jan 13. PMID 25595984
- [Background] Rostami M, Lee A, Frazer AK, Akalu Y, Siddique U, Pearce AJ, Tallent J, Kidgell DJ. Determining the effects of transcranial alternating current stimulation on corticomotor excitability and motor performance: A sham-controlled comparison of four frequencies. Neuroscience. 2025 Mar 5;568:12-26. doi: 10.1016/j.neuroscience.2025.01.016. Epub 2025 Jan 10. PMID 39798837
- [Background] Soleimani G, Kupliki R, Bodurka J, Paulus MP, Ekhtiari H. How structural and functional MRI can inform dual-site tACS parameters: A case study in a clinical population and its pragmatic implications. Brain Stimul. 2022 Mar-Apr;15(2):337-351. doi: 10.1016/j.brs.2022.01.008. Epub 2022 Jan 15. PMID 35042056
- [Background] Chen J, Lin IT, Zhang H, Lin J, Zheng S, Fan M, Zhang J. Reduced cortical thickness, surface area in patients with chronic obstructive pulmonary disease: a surface-based morphometry and neuropsychological study. Brain Imaging Behav. 2016 Jun;10(2):464-76. doi: 10.1007/s11682-015-9403-7. PMID 25986304
- [Background] MacDonald AW 3rd, Cohen JD, Stenger VA, Carter CS. Dissociating the role of the dorsolateral prefrontal and anterior cingulate cortex in cognitive control. Science. 2000 Jun 9;288(5472):1835-8. doi: 10.1126/science.288.5472.1835. PMID 10846167
- [Background] Fried PJ, Santarnecchi E, Antal A, Bartres-Faz D, Bestmann S, Carpenter LL, Celnik P, Edwards D, Farzan F, Fecteau S, George MS, He B, Kim YH, Leocani L, Lisanby SH, Loo C, Luber B, Nitsche MA, Paulus W, Rossi S, Rossini PM, Rothwell J, Sack AT, Thut G, Ugawa Y, Ziemann U, Hallett M, Pascual-Leone A. Training in the practice of noninvasive brain stimulation: Recommendations from an IFCN committee. Clin Neurophysiol. 2021 Mar;132(3):819-837. doi: 10.1016/j.clinph.2020.11.018. Epub 2020 Dec 3. PMID 33549501
- [Background] Amouzadeh F, Sheikh M. Impact of transcranial alternating current stimulation on working memory and selective attention in athletes with attention deficit hyperactivity disorder: randomized controlled trial. Neuroreport. 2022 Dec 14;33(17):756-762. doi: 10.1097/WNR.0000000000001842. Epub 2022 Oct 17. PMID 36250434
- [Background] Gehrman PR, Bartky EJ, Travers C, Lapidus K. A Fully Remote Randomized Trial of Transcranial Alternating Current Stimulation for the Acute Treatment of Major Depressive Disorder. J Clin Psychiatry. 2024 Apr 22;85(2):23m15078. doi: 10.4088/JCP.23m15078. PMID 38696220
- [Background] Hendi NI, El-Samahy M, AboEl-Azm YH, Arar A, Ramadan SI, Zedan EM, et al. Efficacy of Transcranial Alternating Current Stimulation (tACS) in Cognition and Memory in Patients with Mild Cognitive Impairement or Alzheimer's Disease. A Systematic Review and Meta-analysis of Randomized Controlled Trials: Alzheimers Dement. 2025 Jan 9;20(Suppl 6):e087903. doi: 10.1002/alz.087903. eCollection 2024 Dec.; 2025.
- [Background] Tabka O, Sanaa I, Mekki M, Acheche A, Paillard T, Trabelsi Y. Effect of a pulmonary rehabilitation program combined with cognitive training on exercise tolerance and cognitive functions among Tunisian male patients with chronic obstructive pulmonary disease: A randomized controlled trial. Chron Respir Dis. 2023 Jan-Dec;20:14799731231201643. doi: 10.1177/14799731231201643. PMID 37691169
- [Background] Lavoie KL, Sedeno M, Hamilton A, Li PZ, De Sousa D, Troosters T, Maltais F, Bourbeau J. Behavioural interventions targeting physical activity improve psychocognitive outcomes in COPD. ERJ Open Res. 2019 Nov 4;5(4):00013-2019. doi: 10.1183/23120541.00013-2019. eCollection 2019 Oct. PMID 31720294
- [Background] Andrianopoulos V, Gloeckl R, Schneeberger T, Jarosch I, Vogiatzis I, Hume E, Koczulla RA, Kenn K. Benefits of pulmonary rehabilitation in COPD patients with mild cognitive impairment - A pilot study. Respir Med. 2021 Aug-Sep;185:106478. doi: 10.1016/j.rmed.2021.106478. Epub 2021 May 23. PMID 34038843
- [Background] Bonnevie T, Medrinal C, Combret Y, Debeaumont D, Lamia B, Muir JF, Cuvelier A, Prieur G, Gravier FE. Mid-Term Effects of Pulmonary Rehabilitation on Cognitive Function in People with Severe Chronic Obstructive Pulmonary Disease. Int J Chron Obstruct Pulmon Dis. 2020 May 19;15:1111-1121. doi: 10.2147/COPD.S249409. eCollection 2020. PMID 32546999
- [Background] France G, Orme MW, Greening NJ, Steiner MC, Chaplin EJ, Clinch L, Singh SJ. Cognitive function following pulmonary rehabilitation and post-discharge recovery from exacerbation in people with COPD. Respir Med. 2021 Jan;176:106249. doi: 10.1016/j.rmed.2020.106249. Epub 2020 Nov 21. PMID 33253973
- [Background] Turan O, Turan PA, Mirici A. Parameters affecting inhalation therapy adherence in elderly patients with chronic obstructive lung disease and asthma. Geriatr Gerontol Int. 2017 Jun;17(6):999-1005. doi: 10.1111/ggi.12823. Epub 2016 Jul 18. PMID 27426234
- [Background] Dodd JW. Lung disease as a determinant of cognitive decline and dementia. Alzheimers Res Ther. 2015 Mar 21;7(1):32. doi: 10.1186/s13195-015-0116-3. eCollection 2015. PMID 25798202
- [Background] Pelgrim CE, Peterson JD, Gosker HR, Schols AMWJ, van Helvoort A, Garssen J, Folkerts G, Kraneveld AD. Psychological co-morbidities in COPD: Targeting systemic inflammation, a benefit for both? Eur J Pharmacol. 2019 Jan 5;842:99-110. doi: 10.1016/j.ejphar.2018.10.001. Epub 2018 Oct 15. PMID 30336140
- [Background] Yohannes AM, Chen W, Moga AM, Leroi I, Connolly MJ. Cognitive Impairment in Chronic Obstructive Pulmonary Disease and Chronic Heart Failure: A Systematic Review and Meta-analysis of Observational Studies. J Am Med Dir Assoc. 2017 May 1;18(5):451.e1-451.e11. doi: 10.1016/j.jamda.2017.01.014. Epub 2017 Mar 11. PMID 28292570
- [Background] Lindbergh CA, Dishman RK, Miller LS. Functional Disability in Mild Cognitive Impairment: A Systematic Review and Meta-Analysis. Neuropsychol Rev. 2016 Jun;26(2):129-59. doi: 10.1007/s11065-016-9321-5. Epub 2016 Jul 8. PMID 27393566
- [Background] Torres-Sanchez I, Rodriguez-Alzueta E, Cabrera-Martos I, Lopez-Torres I, Moreno-Ramirez MP, Valenza MC. Cognitive impairment in COPD: a systematic review. J Bras Pneumol. 2015 Mar-Apr;41(2):182-90. doi: 10.1590/S1806-37132015000004424. Epub 2015 Apr 18. PMID 25909154
- [Background] Dhakal A, Bobrin BD. Cognitive Deficits. StatPearls. Treasure Island (FL) ineligible companies. Disclosure: Bradford Bobrin declares no relevant financial relationships with ineligible companies.: StatPearls Publishing Copyright © 2023, StatPearls Publishing LLC.; 2023.
- [Background] Dodd JW, Getov SV, Jones PW. Cognitive function in COPD. Eur Respir J. 2010 Apr;35(4):913-22. doi: 10.1183/09031936.00125109. PMID 20356988
- [Background] Ranzini L, Schiavi M, Pierobon A, Granata N, Giardini A. From Mild Cognitive Impairment (MCI) to Dementia in Chronic Obstructive Pulmonary Disease. Implications for Clinical Practice and Disease Management: A Mini-Review. Front Psychol. 2020 Feb 28;11:337. doi: 10.3389/fpsyg.2020.00337. eCollection 2020. PMID 32184750
- [Background] Samareh Fekri M, Hashemi-Bajgani SM, Naghibzadeh-Tahami A, Arabnejad F. Cognitive Impairment among Patients with Chronic Obstructive Pulmonary Disease Compared to Normal Individuals. Tanaffos. 2017;16(1):34-39. PMID 28638422

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-07-25): https://cdn.clinicaltrials.gov/large-docs/69/NCT07332169/Prot_SAP_000.pdf
  • Informed Consent Form (2025-07-25): https://cdn.clinicaltrials.gov/large-docs/69/NCT07332169/ICF_001.pdf